CLINICAL TRIAL: NCT02711384
Title: Minimum Alveolar Concentration of Sevoflurane for Maintaining BIS Below 50 in Patients Undergoing Coronary Artery Bypass Grafting During Normothermic Cardiopulmonary Bypass Phase.
Brief Title: MACBIS50 in Patients Undergoing CAG During Normothermic CPB Phase.
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Carlos Gustavo dos Santos Silva, MD, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 4555
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Coronary Disease; Coronary Artery Disease
Keywords: Sevoflurane; Coronary artery bypass grafting; Cardiopulmonary bypass; Inhalation anesthesia; MACBIS50
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: We determined the minimum alveolar concentration (MAC) of sevoflurane for maintaining bispectral index (BIS) below 50 (MACBIS50) in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase. Method: Fifteen patients, American Society of Anestesiology physical status III or IV, aged 40-70, undergoing elective coronary artery bypass grafting, were enrolled in our study. The predetermined target end-tidal sevoflurane concentration was maintained for at least ten minutes during normothermic cardiopulmonary bypass phase. BIS values were then recorded at an interval of 10 s for 1 min. The dial settings were adjusted to attain an end-tidal sevoflurane concentration of 1% in the first patient. If a given patient had an average BIS of < 50, the sevoflurane concentration was reduced by 0.1% in the subsequent patient, whereas if a given patient had a BIS ≥ 50, the sevoflurane concentration was increased by 0.1% in the next patient. MACBIS50 was calculated using the midpoint concentration of patients involving a crossover according to the up-down method. Average of the crossover midpoints in each pair defined effective dose 50. Data were also analyzed by a logistic regression test to obtain the probability of BIS < 50 versus end-tidal sevoflurane concentration. Result: MACBIS50 of sevoflurane was 0,82% (95% confidence intervals: 0,47-1,16) in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase. Conclusion: MACBIS50 determined in this study was 15% lower compared to MACBIS50 in middle-aged adults after tracheal intubation.

DETAILED DESCRIPTION:
Minimum alveolar concentration (MAC) is defined as the minimum alveolar concentration at sea level of inhaled anaesthetic required to prevent apparently purposeful movement in 50% of patients in response to surgical incision1,2. A similar approach to the one described to ascertain MAC has been used to determine the potency of inhaled anaesthetics for other desirable clinical end-points of general anaesthesia, such as to maintain bispectral index (BIS) below 50 (MACBIS50). Therefore, MACBIS50 is defined as the minimum alveolar concentration of inhaled anaesthetic for maintaining BIS below 50 in 50% of patients. MACBIS50 was determined in different age groups and clinical conditions of patients, but not in cardiac surgery3-5.

This study aims to determine the minimum alveolar concentration of sevoflurane for maintaining bispectral index below 50 in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase.

Methods After obtaining approval from the institutional ethics committee and written informed consent, fifteen patients, American Society of Anestesiology physical status III or IV, aged 40-70, undergoing elective coronary artery bypass grafting, were enrolled in our study. Exclusion criteria included history of psychiatric or neurological diseases, drug abuse or medications that affect the central nervous system, pregnancy, combined surgeries, reoperation in cardiac surgery, emergency procedures and neuraxial block.

No premedication was given. Intraoperative monitoring consisted of a five-lead ECG, pulse oximetry, gas analyzer, bladder catheterization, invasive arterial pressure in the radial artery, esophageal thermometer, central venous catheter inserted through the subclavian vein, transesophageal echocardiography (when indicated), train-of-four monitoring (TOF) and BIS (BIS Vista™; Covidien). Breath-by-breath inspired/end-tidal sevoflurane and carbon dioxide (CO2) concentrations were measured with a multigas analyzer and it was calibrated before each experiment. The anaesthetic system used was a semi-closed system (Primus® - Draeger).

Anesthesia was induced with sevoflurane in 6 L.min-1 oxygen using the incremental increase technique via a face mask until the loss of consciousness and BIS value between 40-60. After then sufentanil (0.5 µg.kg-1) and pancuronium (0.1 µg.kg-1) were given and assisted ventilation was started. The T4/T1 ratio was measured using the TOF every minute until orotracheal intubation. The patient was intubated with the following parameters: BIS value between 40-60 and TOF = 0. Mechanical ventilation was initiated using controlled-volume mode (tidal volume of 6 mL.kg-1, ventilatory frequency of 12-15 bpm, PEEP of 5 mmHg and minute ventilation adjusted to maintain end-tidal carbon dioxide tension with the range of 35-40 mmHg). Neuromuscular block was maintained under deep block (TOF = 0 and PTC ≥ 1) using pancuronium up to one hour before the end of the procedure. Anesthesia was maintained using sufentanil (1 µg.kg-1 before the surgical incision) and up to 1 MAC of the end-tidal sevoflurane to maintain a BIS between 40-60. Continuous norepinephrine infusion was started if the mean arterial pressure was less than 60 mmHg.

Patients were anticoagulated with heparin (400 U.kg-1) before insertion of the aortic cannula. Anesthesia was maintained using up to 1 MAC of the end-tidal sevoflurane to maintain a BIS between 40-60 during cardiopulmonary bypass (CPB), measured by the gas analyzer positioned after the membrane oxygenator of the CPB circuit.

The predetermined target end-tidal sevoflurane concentration was maintained for at least ten minutes during normothermic cardiopulmonary bypass phase (36,5 degrees celsius). BIS values were then recorded at an interval of 10 seconds for 1 min. The dial settings were adjusted to attain an end-tidal sevoflurane concentration of 1% in the first patient. If a given patient had an average BIS of < 50, the sevoflurane concentration was reduced by 0.1% in the subsequent patient, whereas if a given patient had a BIS ≥ 50, the sevoflurane concentration was increased by 0.1% in the next patient.

EEG data were continuously observed by a monitor. The impedance of each electrode was maintained at < 2 kΩ. The smoothing window was set at 15s, which was used for interpreting the data.

Statistics Patient characteristic and intraoperative data were collected and presented as mean ± standard deviation. The Dixon's up-and-down method needs six pairs of failure-success for statistical analysis. MACBIS50 was calculated using the midpoint concentration of patients involving a crossover (BIS < or ≥ 50) according to the up-down method. Average of the crossover midpoints in each pair defined effective dose (ED50). The up-and-down sequences were also analyzed by the probit test, which enabled us to derive the sevoflurane concentration for maintaining BIS of 50, with 95% confidence limits of the mean. Data were also analyzed by a logistic regression test to obtain the probability of BIS < 50 versus end-tidal sevoflurane concentration, the maximum likelihood estimators of the model variables, and a goodness of fit.

Results A total of fifteen patients were recruited for this study (figure 1). The patient characteristics and intraoperative data are shown in Table 1. Sequences of individual patients according to up-down method are shown in Figure 2. MACBIS50 of sevoflurane was 0,82% (95% confidence intervals: 0,47-1,16) in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase. MACBIS50 value estimated with probit analysis (Figure 3) was 0,73% (95% confidence intervals: 0,45-1,00), which was similar to that derived from up-down method. Corresponding ED95 values (minimum concentration of sevoflurane required for maintaining BIS value < 50 in 95% subjects) was 1,39 (95% confidence intervals: 0,42-2,37).

No patient had dysrhythmia, hypotension or bradycardia at the moment of BIS measurement. Dobutamine (0.5 µg.kg-1.min-1) was administered for all patients during normothermic cardiopulmonary bypass phase.

Discussion This study showed that MACBIS50 of sevoflurane was calculated to be 0,82% (95% confidence intervals: 0,47-1,16) in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase. This value was 15% lower compared to MACBIS50 in middle-aged adults after tracheal intubation (0.97%; 95% confidence intervals: 0.89- 1.05)3. Matsuura et al. showed that MACBIS50 of sevoflurane in young, middle-aged, and elderly patients was 1.28% (1.24-1.32), 0.97% (0.89-1.05), and 0.87% (0.84-0.90), respectively. The MACBIS50 was significantly higher in young patients and significantly lower in elderly patients than those in middle-aged patients3.

Regarding our study, decreased MACBIS50 may be related to some factors such as hemodilution and use of opioids during surgery. Administration of 5% isotonic dextrose reduced both cerebrospinal fluid sodium and osmolality. This dilution of cerebrospinal fluid sodium was associated with a reduction in MAC. That correlation did not occur with other solutions6. Therefore, perhaps the hemodilution of the CPB circuit with 0.9% saline solution did not interfere with the determination of MACBIS50 of sevoflurane in our study. In the other hand, MAC consistently decreased with a decrease in cerebrospinal fluid sodium6. In this way, it may have been a limiting factor for the determination of MACBIS50 of sevoflurane in our study.

Studies using loading doses followed by infusions of sufentanil administered until just before CPB have demonstrated a decrease in sufentanil concentrations of 30-55% on commencing CPB7,8. Concentrations are stable during hypothermic CPB and then increase on rewarming, indicating that relatively large amounts of sufentanil are sequestered in the tissues during hypothermic CPB and released during rewarming. Immediately after CPB, sufentanil concentrations approach pre-CPB values. The increase in sufentanil concentration on rewarming implies that binding of sufentanil to the CPB circuit is unlikely, and the stability of the concentrations during CPB suggests that metabolism and excretion do not occur during this period8.

In the other hand, studies on infusions of sufentanil throughout CPB have demonstrated a decrease of less than 20 % in total sufentanil concentration on commencing CPB9. There was no correlation between sufentanil concentration and either total protein or albumin concentrations, which both decreased by a greater percentage. The relatively small decrease in sufentanil concentration is explained by rapid redistribution of free drug from the tissues to the blood. Sufentanil has a large volume of distribution and hence the change in volume as a result of the prime is small8.

In addition to the pharmacokinetic characteristics of sufentanil in CPB, there is interaction between opioids and inhaled anesthetics. Sufentanil produces similar reduction in isoflurane MAC, with an initial steep reduction at lower concentrations and a plateau effect at higher concentrations10. We used a total dose of 1.5 µg.kg-1 of sufentanil (0.5 µg.kg-1 for anesthetic induction and 1.0 µg.kg-1 before the surgical incision). Therefore, the pharmacokinetic characteristics of sufentanil in CPB associated with the interaction between opioids and inhaled anesthetics may justify a lower MACBIS50 in the population of our study.

Nussmeier et al. showed that washin of isoflurane appeared to occur more slowly during CPB than during administration via the lungs in normothermic patients, presumably because hypothermia increases tissue capacity. During rewarming, washout appeared to occur as rapidly as from the lungs of normothermic patients11.

We used BIS value below 50 as an index of the depth of anaesthesia. We considered the end-tidal concentrations to maintain BIS below 50 as an appropriate concentration to achieve hypnotic responses. As supportive evidence, this value has been used previously by other researchers3,12. We did not investigate other BIS values such as 40 or 60. Assessment of the relationships between anaesthetic concentrations and a variety of BIS values would warrant further study, but BIS value below 50 is supposed to play a role as an index indicative of adequate depth of anaesthesia. However, BIS values more than 60 would entail a risk of awareness during procedure13.

MAC increased significantly only during ephedrine infusion. Mephentermine, phenylephrine, metaraminol, methoxamine, noradrenaline and adrenaline did not change MAC14. However, no studies on the effects of dobutamine infusion and MAC of inhaled anesthetics.

In summary, our study is a pioneer in determining MACBIS50 in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase. Therefore, further studies to determine the MACBIS50 of sevoflurane in different age groups should be developed in the context of coronary artery bypass grafting and other cardiac procedures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anestesiology physical status III or IV;
* Aged 40-70;
* Undergoing elective coronary artery bypass grafting.

Exclusion Criteria:

* History of psychiatric or neurological diseases;
* Drug abuse or medications that affect the central nervous system;
* Pregnancy;
* Combined surgeries;
* Reoperation in cardiac surgery;
* Emergency procedures;
* Neuraxial blockade.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Society of Anestesiology physical status III or IV, aged 40-70, undergoing elective coronary artery bypass grafting
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
MACBIS50 in patients undergoing CAG during normothermic CPB phase. | 1 year
  To determine the minimum alveolar concentration of sevoflurane for maintaining bispectral index below 50 in patients undergoing coronary artery bypass grafting during normothermic cardiopulmonary bypass phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No